CLINICAL TRIAL: NCT03895879
Title: Concentration-guided Dose Reduction Versus Standard Dosing in Tocilizumab-treated Rheumatoid Arthritis Patients: a Randomised, Multicenter, Non-inferiority Trial (TODORA)
Brief Title: Use of Tocilizumab Drug Levels to Optimize Treatment in RA
Acronym: TODORA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Reade Rheumatology Research Institute (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TODORA; 2018-004605-57 (EudraCT Number); NL68462.029.19 (Other: Medical Ethical Committee VUmc, Amsterdam)
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Tocilizumab; Therapeutic Drug Monitoring; Drug level; Dose reduction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Patients with tocilizumab trough concentrations above 15 mg/L will be randomly assigned to dose reduction by increasing their dosing interval from once every week to once every two weeks, or to continuation of the standard dose. All patients with concentrations below 15 mg/L during the first study visit will not be randomized and all continue standard treatment.
Who Masked: Outcomes Assessor
Masking Description: During every study visit the joints of all patients will be examined for pain and swelling by a blinded nurse or physician. The number of painful and swollen joints will be used to calculate the DAS28 score, the primary outcome of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention (Experimental): Tocilizumab administered every 2 weeks
  Interventions: Drug: Tocilizumab
- Control (Active Comparator): Tocilizumab administered every week
  Interventions: Drug: Tocilizumab
- Standard dose (screening < 15 mg/L) (Active Comparator): Tocilizumab administered every week
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab sc (162 mg) once every 2 weeks
  Arms: Intervention
Drug: Tocilizumab — Tocilizumab sc (162 mg) once every week
  Arms: Control; Standard dose (screening < 15 mg/L)

SUMMARY:
Tocilizumab concentrations above 1 mg/L are likely to be sufficient for normalizing C-reactive protein (CRP) production in patients with rheumatoid arthritis (RA). In practice, however, a large variability in the concentrations of tocilizumab is found, and a large proportion of patients treated with tocilizumab subcutaneously (sc) have concentrations far above 1 mg/L. These patients can probably lower their doses without losing clinical response.

A 52 weeks non-inferiority, multicenter, randomized controlled study will be performed to investigate whether patients with RA with serum trough concentrations of tocilizumab higher than 15 mg/L can increase their dosing interval to every two weeks without losing clinical response. Patients with relatively high trough concentrations will be randomly assigned to continuation of the standard dose or to increase dosing interval to every two weeks. The main objective is to investigate the difference in mean time weighted Disease Activity Score in 28 joints, including erythrocyte sedimentation rate (DAS28-ESR) between the two groups after 28 weeks. It is expected that patients with relatively high trough concentrations can safely increase their dosing interval without losing response.

DETAILED DESCRIPTION:
Tocilizumab is a humanized monoclonal antibody targeting the IL-6 receptor (IL-6R). It has proven to be effective in reducing inflammation and symptoms in rheumatoid arthritis (RA). The registered standard dose of tocilizumab subcutaneously (sc) is 162 mg weekly for every patient. All patients diagnosed with RA and treated with tocilizumab sc receive the same dose, so treatment with expensive biologicals is currently based on a 'one size fits all' approach. Because of the large inter-individual variability in the pharmacokinetics of tocilizumab this standard dose results in a wide range of serum concentrations. In the search to optimize the dose for individual patients it was demonstrated that serum levels of 1 mg/L of tocilizumab are adequate to block the IL-6 receptor systemically, as indicated by a reduction in CRP levels in patients with these low trough concentrations. Therefore, a substantial proportion of patients is likely to be overexposed to tocilizumab. This overtreatment is a waste of health care resources and might be associated with an increased risk of adverse events, mainly infections.

We believe that overexposure can be reduced effectively by making use of the drug concentrations found in the serum of individual patients. Our hypothesis is therefore that reducing the dose in the setting of therapeutic drug monitoring (TDM) does not affect clinical disease activity and safety, while it will reduce costs.

Based on previous studies we believe that a concentration around 5 mg/L is sufficient to reach the maximal treatment effect. Therefore tapering strategy was developed aiming for serum concentrations around 5 mg/L. Monte Carlo modelling was performed to determine the cut-off concentration for interval prolongation to be used in this study. Simulations were performed and it was found that patients with trough concentrations above 15 mg/L can safely prolong their dosing interval, as this will result in levels around 5 mg/L in the majority of patients.

This study is a 52 weeks randomised, multicenter, non-inferiority trial in rheumatoid arthritis patients treated with subcutaneous tocilizumab 162 mg weekly for at least the previous 6 months. After informed consent is obtained during the baseline visit, blood will be drawn to measure drug trough concentrations. Patients with a tocilizumab concentration above 15 mg/L will be randomly assigned to dose reduction by increasing their dosing-interval from once every week to once every two weeks, or to continuation of their tocilizumab dose (standard dose). After randomization, patients are followed for a period of 52 weeks. Data regarding disease status and functioning will be collected during the baseline visit, and 12, 28, 40, and 52 weeks thereafter. Blood will also be drawn from the patients during these visits. All patients with concentrations below 15 mg/L during the first study visit will not be randomized and all continue standard treatment. Only one follow-up visit, after 52 weeks, will be performed in this group of patients.

Patients can also choose to participate in a sub-study where the finger prick developed by Sanquin (Amsterdam) will be validated to measure tocilizumab drug levels. This part of the study will comprise performing three finger pricks. These finger pricks will be performed during the visit at week 12 with the help of a nurse, and at home during the two weeks after this visit.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to the American College of Rheumatology (ACR) 1987 or 2010 criteria;
* Current use of subcutaneous tocilizumab 162 mg weekly, for at least the previous 6 months;
* The treating rheumatologist is convinced of the benefit of tocilizumab continuation;
* Written informed consent.

Exclusion Criteria:

* A scheduled surgery in the next 52 weeks or other pre-planned reasons for treatment discontinuation;
* Changes in the treatment with glucocorticoids and DMARDs such as methotrexate in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
DAS28-ESR | 28 weeks
  The difference in mean time weighted DAS28 after 28 weeks between patients undergoing concentration-guided dose reduction or standard dosing.

SECONDARY OUTCOMES:
DAS28-ESR | 52 weeks
  The difference in mean time weighted DAS28 after 52 weeks between patients undergoing concentration-guided dose reduction or standard dosing.
Clinical Disease Activity Index (CDAI) | 28 and 52 weeks
  The difference in CDAI-score after 28 and 52 weeks between the patients undergoing concentration-guided dose reduction or standard dosing.
Simple Disease Activity Index (SDAI) | 28 and 52 weeks
  The difference in SDAI-score after 28 and 52 weeks between the patients undergoing concentration-guided dose reduction or standard dosing.
Health Assessment Questionnaire (HAQ) | 28 and 52 weeks
  The difference in HAQ-score after 28 and 52 weeks between the patients undergoing concentration-guided dose reduction or standard dosing.
Direct medical costs of TDM | 52 weeks
  The difference in direct medical costs of TDM compared to the standard treatment regimen.
Number of flares | 28 and 52 weeks
  The difference in number of flares at 28 and 52 weeks between patients undergoing concentration-guided dose reduction or standard dosing.
Number and severity of adverse events | 28 and 52 weeks
  The difference in number and severity of adverse events at 28 and 52 weeks between patients undergoing concentration-guided dose reduction or standard dosing.
Drug level | 52 weeks
  The difference in drug levels in the intervention group between week 0 and 52.
Patient perspective towards therapeutic drug monitoring | 52 weeks
  A questionnaire will be used to evaluate the perspective of patients towards therapeutic drug monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Wolbink, MD, PhD, Principal Investigator — Reade Rheumatology Research Institute
Locations (1):
- Reade Rheumatology Research Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
To avoid duplication of research, the data gathered in this study will be shared once all desirable data analysis have been performed and the results are published.
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the final publication from the study is published the data will be shared.
Access Criteria: Researchers with demonstrable interest in autoimmunity, biologicals, or TDM can contact the investigators of the trial if they are interested in gaining access to the data. Depending on their research objectives the data will be shared.

REFERENCES:
- [Background] Kneepkens EL, van den Oever I, Plasencia CH, Pascual-Salcedo D, de Vries A, Hart M, Nurmohamed MT, Balsa A, Rispens T, Wolbink G. Serum tocilizumab trough concentration can be used to monitor systemic IL-6 receptor blockade in patients with rheumatoid arthritis: a prospective observational cohort study. Scand J Rheumatol. 2017 Mar;46(2):87-94. doi: 10.1080/03009742.2016.1183039. Epub 2016 Jul 20. PMID 27440258
- [Background] l'Ami MJ, Krieckaert CL, Nurmohamed MT, van Vollenhoven RF, Rispens T, Boers M, Wolbink GJ. Successful reduction of overexposure in patients with rheumatoid arthritis with high serum adalimumab concentrations: an open-label, non-inferiority, randomised clinical trial. Ann Rheum Dis. 2018 Apr;77(4):484-487. doi: 10.1136/annrheumdis-2017-211781. Epub 2017 Sep 22. PMID 28939629
- [Background] Frey N, Grange S, Woodworth T. Population pharmacokinetic analysis of tocilizumab in patients with rheumatoid arthritis. J Clin Pharmacol. 2010 Jul;50(7):754-66. doi: 10.1177/0091270009350623. Epub 2010 Jan 23. PMID 20097931
- [Background] Bastida C, Ruiz-Esquide V, Pascal M, de Vries Schultink AHM, Yague J, Sanmarti R, Huitema ADR, Soy D. Fixed dosing of intravenous tocilizumab in rheumatoid arthritis. Results from a population pharmacokinetic analysis. Br J Clin Pharmacol. 2018 Apr;84(4):716-725. doi: 10.1111/bcp.13500. Epub 2018 Feb 7. PMID 29314183